CLINICAL TRIAL: NCT07205003
Title: Evaluation of the Link Between Carotid Arterial Wall Viscosity and Major Neurocognitive Disorders of Vascular Origin or Linked to Alzheimer's Disease
Brief Title: Evaluation of the Link Between Carotid Arterial Wall Viscosity and Major Neurocognitive Disorders
Acronym: VISCOG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/021/OB; 2021-A00291-40 (Other: ANSM)
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Neurocognitive Disorders; Alzheimer's Disease
Keywords: carotid arterial wall viscosity
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — In this context, an additional 4 mL EDTA tube will be collected to evaluate Alzheimer's disease biomarkers. This sample will be centrifuged to obtain six 150 μL aliquots and one 1 mL aliquot, which will then be stored at -80°C. The SIMOA® technique will allow the following Alzheimer's markers to be measured: Aβ1-40 and 1-42, Tau (the 3 included in the Neurology 3-Plex A kit), phosphoTau 181 and 231.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of carotid wall viscosity in patients with vascular dementia — Carotid wall viscosity will be assessed by simultaneous and continuous measurement by 2 operators of local pressure and diameter at the level of the right and left carotids by coupling echotracking (Vevo 3100®) with applanation tonometry (Millar®). 3 successive measurements will be carried out. These measurements will establish the diameter-pressure relationship and its analysis will allow the calculation of wall viscosity by measuring the area under the curve of this relationship during the cardiac cycle.
Diagnostic Test: Assessment of carotid wall viscosity in patients with Alzheimer's disease — Carotid wall viscosity will be assessed by simultaneous and continuous measurement by 2 operators of local pressure and diameter at the level of the right and left carotids by coupling echotracking (Vevo 3100®) with applanation tonometry (Millar®). 3 successive measurements will be carried out. These measurements will establish the diameter-pressure relationship and its analysis will allow the calculation of wall viscosity by measuring the area under the curve of this relationship during the cardiac cycle.
Diagnostic Test: Assessment of carotid wall viscosity in patients not presenting dementia. — Carotid wall viscosity will be assessed by simultaneous and continuous measurement by 2 operators of local pressure and diameter at the level of the right and left carotids by coupling echotracking (Vevo 3100®) with applanation tonometry (Millar®). 3 successive measurements will be carried out. These measurements will establish the diameter-pressure relationship and its analysis will allow the calculation of wall viscosity by measuring the area under the curve of this relationship during the cardiac cycle.

SUMMARY:
The mechanical behavior of conductance arteries is viscoelastic. While the elastic component has been extensively studied, the viscous component has often been neglected for methodological reasons and also because it was considered weak.

Unlike a purely elastic solid, which exhibits instantaneous deformation/relaxation upon application/discontinuation of a force, a viscoelastic solid is characterized, from a mechanical point of view, by a delay between the application or discontinuation of the force and deformation. Thus, at the arterial level, the elasticity of the arterial wall allows the internal diameter to increase proportionally to the blood pressure during systole. The viscous component will induce a delay in diameter restoration, resulting in a larger diameter at each pressure level during the diastolic phase compared to the systolic phase. This results in a shift between the systolic and diastolic curves of the pressure-diameter relationship, creating a hysteresis loop. From a thermodynamic point of view, while a purely elastic material fully restores the energy stored during the loading phase, viscoelastic arteries will incompletely restore this energy. Thus, the surface of the hysteresis loop reflects the energy dissipated during each cardiac cycle (WV), and the area under the loading phase curve represents the energy stored by the arterial wall (WE) during the latter. Thus, arterial wall viscosity (APV) can be expressed either as the absolute value of WV or as a function of the stored energy (WV/WE). Physiologically, this energy loss is low. Its increase could be accompanied by excessive energy dissipation, leading to increased cardiac work and cardio-circulatory decoupling. Conversely, low parietal viscosity could lead to damage to peripheral organs by excessive transmission of pulsatile energy to the periphery due to lack of damping.

DETAILED DESCRIPTION:
Preliminary work in the laboratories has highlighted the role of vaso-relaxing endothelial factors and smooth muscle tone in the regulation of the Arterial Pulse Rate (APR) of the radial artery in the basal and stimulated state and the alteration of this stimulated regulation during Arterial Hypertension (AH). Furthermore, a decrease in relative carotid APR in middle-aged subjects compared to young subjects, and an increase in carotid APR in diabetic patients has been found in unpublished results. The link between aortic arterial stiffness and the existence of vascular dementia but also Alzheimer's is strongly suggested. Indeed, the increase in arterial stiffness could be responsible for an increase in pulsatility transmitted to the brain, participating in the accumulation of beta amyloid proteins. A probable inflammatory and oxidative stress component could also have an added deleterious role through the production of free radicals. Thus, previous studies have shown the existence of a link between arterial stiffness and the presence of leukoaraiosis, lacunae, microbleeds but also with brain volume and the progression of cerebral atrophy. These repercussions on the cerebral parenchyma are visible on MRI.

A link has also been suggested between increased arterial stiffness and impaired cognitive function (as demonstrated by neurocognitive tests) or the presence of markers of small vessel damage in neuroimaging (microbleeds, lacunae, leukoaraiosis). One hypothesis to explain this link is that arterial stiffness promotes impaired hippocampal microcirculation. Other studies have shown that carotid-femoral pressure wave velocity (CFV), a marker of large arterial stiffness, was higher in populations with Alzheimer's disease and vascular dementia than in older populations without cognitive impairment or with minor neurocognitive impairment.

However, no studies have evaluated the link between baseline VPA and vascular dementia or Alzheimer's disease.

Our study suggests that carotid VPA is associated with increased cerebrovascular injury, impaired cognitive testing, and the diagnosis of vascular dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age over 70
* Memory consultation consultant (neurology or geriatrics)
* Brain MRI less than one year old or planned as part of the cognitive assessment performed.
* Patient diagnosed with Alzheimer's disease according to DSM-5 criteria or vascular dementia according to DSM-5 criteria, or presenting a memory complaint without evidence of a dementia-related condition.
* No objection from the patient or their caregiver.
* Patient covered by a health insurance plan

Exclusion Criteria:

* Known unilateral or bilateral carotid stenosis or history of carotid surgery
* Permanent CA/AF
* Patient presenting with confusion
* Known psychiatric illness (severe depression, psychosis, etc.)
* Non-vascular, non-Alzheimer's dementia (e.g., Lewy Body Dementia, Parkinsonian Dementia, Progressive Supranuclear Palsy)
* Refusal to participate
* MMS less than or equal to 10
* Contraindication to performing an MRI
* Any acute decompensated pathology
* Patient under guardianship or curatorship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 140 sujets dont 55 sujets avec démence vasculaire et 55 avec une démence de type maladie d'Alzheimer et 30 avec plainte mnésique sans troubles neurocognitifs.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the difference in relative arterial wall viscosity value of the common carotid artery of patients with vascular dementia compared to that of patients with Alzheimer's disease | enrollment visit
  Carotid wall viscosity will be assessed using a method developed in the pharmacology department, involving simultaneous and continuous measurement by two operators of local pressure and diameter at the right and left carotid arteries, combining echotracking (Vevo 3100®) with applanation tonometry (Millar®). Three successive measurements will be performed. These measurements will establish the diameter-pressure relationship, and their analysis will allow calculation of wall viscosity by measuring the area under the curve of this relationship during the cardiac cycle. The primary outcome measure will be the difference in carotid arterial wall viscosity between the two groups of subjects; it will be studied by analysis of variance (ANOVA).
Evaluation of the difference in relative arterial wall viscosity value of the common carotid artery of patients with vascular dementia compared to that of patients not presenting dementia | enrollment visit
  Carotid wall viscosity will be assessed using a method developed in the pharmacology department, involving simultaneous and continuous measurement by two operators of local pressure and diameter at the right and left carotid arteries, combining echotracking (Vevo 3100®) with applanation tonometry (Millar®). Three successive measurements will be performed. These measurements will establish the diameter-pressure relationship, and their analysis will allow calculation of wall viscosity by measuring the area under the curve of this relationship during the cardiac cycle. The primary outcome measure will be the difference in carotid arterial wall viscosity between the two groups of subjects; it will be studied by analysis of variance (ANOVA).

SECONDARY OUTCOMES:
Evaluation of the link between arterial parietal viscosity of the common carotid artery and the intensity of cerebral vascular | enrollment visit
  Establishment of the correlation between the relative arterial parietal viscosity value of the common carotid artery and the intensity of lesions in MRI (Fazekas Classification). The Fazekas classification is a system used in neurology and neuroradiology to assess and grade the severity of cerebral white matter lesions observed on MRI. (Low grades (0-1): Changes are often age-related and without major symptoms. High grades (2-3): Indicate more severe impairment, associated with a greater risk of cognitive impairment)
Study of the link between arterial parietal viscosity of the common carotid artery and the severity of cognitive impairment (MMSE) | enrollment visit
  Measurement of the correlation between the relative arterial parietal viscosity value and cognitive performance score MMSE. This is a short, standardized test used to assess overall cognitive function (score 27-30 Normal cognitive function; score 21-26 Mild cognitive impairment; score 10-20 Moderate impairment; score <10 Severe impairment)
Study of the link between arterial parietal viscosity of the common carotid artery and the severity of cognitive impairment (Gröber test) | enrollment visit
  Measurement of the correlation between the relative arterial parietal viscosity value and cognitive performance score Gröber test. This neuropsychological test assesses verbal episodic memory, that is, the ability to memorize and recall verbal information. This score quantifies an individual's cognitive performance on the Gröber Verbal Memory Test. The score reflects the individual's ability to learn, retain, and recall a list of words presented orally. This assesses the quality of short-term and long-term memory. (A high score indicates good verbal episodic memory. A low score may indicate memory impairment, such as in Alzheimer's disease, other forms of dementia, or following a traumatic brain injury.)
Study of the link between arterial parietal viscosity of the common carotid artery and the severity of cognitive impairment (verbal fluency) | enrollment visit
  Measurement of the correlation between the relative arterial parietal viscosity value and cognitive performance score verbal fluency. Verbal fluency assesses cognitive ability, measuring how easily a person can produce words in response to a given instruction, often within a limited time. (High score = good word production ability, preserved cognitive functioning. Low score = lexical difficulties, executive dysfunction, or cognitive slowing.)
Study of the link between arterial parietal viscosity of the common carotid artery and the severity of cognitive impairment (cognitive performance score (BREF)) | enrollment visit
  Measurement of the correlation between the relative arterial parietal viscosity value and cognitive performance score (BREF). The Cognitive Performance Score (BREF) is a standardized measure used to assess a person's overall cognitive functioning. The score is given on a scale where a lower score indicates better cognitive performance, and a higher score reflects a more marked deficit.
Study of the link between arterial parietal viscosity of the common carotid artery and the severity of cognitive impairment (score oral naming score (DO80)) | enrollment visit
  Measurement of the correlation between the relative arterial parietal viscosity value and cognitive performance score oral naming score (DO80) carry out by assessing the ability to find and produce the exact name of an object (lexical denomination).
Study of the link between arterial parietal viscosity of the common carotid artery and the severity of cognitive impairment (number of successful gestural praxis) | enrollment visit
  Measurement of the correlation between the relative arterial parietal viscosity value and the number of successful gestural praxis perform by measuring the ability to perform voluntary, coordinated and purposeful gestures, particularly learned or symbolic gestures (such as greeting, using a tool, making a sign)..
link between arterial stiffness (carotid and aortic) and the intensity of cerebral vascular lesions in MRI | Enrollment visit
  Measurement of the correlation between segmental arterial stiffness of the common carotid artery (modulus, distensibility) and the intensity of cerebral vascular lesions in MRI.
Link between arterial stiffness (carotid and aortic) and the intensity of cerebral vascular lesions in MRI as well as with the severity of cognitive impairment | enrollment visit
  Measurement of the correlation between segmental arterial stiffness of the common carotid artery (modulus, distensibility) and severity of cognitive impairment

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.